CLINICAL TRIAL: NCT04684927
Title: Post-approval Study to Evaluate the Continued Safety and Efficacy of the MID-C System 5 Years Post-implantation in Adolescent Idiopathic Scoliosis (AIS)
Brief Title: PMS Evaluation of Safety and Efficacy of the MID-C System 5 Years Post-implantation in AIS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: project not initiated
Sponsor: Apifix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MID-C AIS 06-19
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Intervention Model Description: The study is a prospective, single arm, non-randomized, new enrollment cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MID-C treatment (Experimental): Follow-up measurements during 5 years post MIC-C system implantationin order to evaluate safety and efficacy parameters.
  Interventions: Device: MID-C System -Minimal invasive deformity correction system for the treatment of AIS

INTERVENTIONS:
Device: MID-C System -Minimal invasive deformity correction system for the treatment of AIS — A 5 years follow-up will be performed for all patients who underwent AIS repair surgery using the MID-C System. The follow-up in order to assess safety and efficacy measurments. Eligible Patients will be followed and assessed at the following time points: Immediate Post-op up to 6 weeks, 6 months, 12 months, and then annually out to 5 years post-implantation.
  During the study, the following rating scales and assessments will be conducted to assess the probable benefit and safety of the treatment: Physical exam,X-rays,Cobb angle measurements,Adverse Events (AEs) and Scoliosis research society (SRS-22) questionnaire: The questionnaire is commonly used to assess health related quality of life in children with AIS.

SUMMARY:
The ApiFix MID-C System is a unidirectional expandable rod, designed to be connected unilaterally to the spine via 2 anchor points on the concave side of a scoliotic deformity above and below the apex of the major curvature to treat adolescent idiopathic scoliosis. The MID-C System is designed to act as an internal brace. A total of 10 patients, who are planned to undrego the MID-C System implantation procedure will be enrolled for the study. A 5 years follow-up post surgery will be performed for these patients in order to evaluate the long term safety and efficacy of the MID-C System.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent Idiopathic Scoliosis classified as Lenke Type 1 or Type 5 curves; 2.

* Patients with Risser stage 0-1, primary Cobb angle between 35-50 degrees (inclusive), or
* Patients with Risser stage 0-1 and good brace compliant but curve progression above 6°, or
* Patients with Risser stage 0-1 that are non-compliant with brace treatment and primary Cobb angle between 30-50 degrees or
* Patients with Risser stage 2, primary Cobb angle between 40-50 degrees (inclusive) 3. Flexible curve that that reduces to ≤ 30 degrees on lateral side-bending radiographs or as evident by traction x-ray; 4. Kyphosis angles of ≤ 45 degrees measured from T5 to T12; 5. Appropriate candidate for posterior surgical approach; 6. Patient has good general health; 7. Patient has no known hypersensitivity or allergies to titanium; 8. Patient's guardian signs a written informed consent form (ICF).

Exclusion Criteria:

1. Any type of non-idiopathic scoliosis;
2. Any main thoracic deformity that includes vertebral levels and cranial including to T2;
3. Cumulative vertebral wedging over the apex of the curve>15º
4. Known history of existing malignancy, or any systemic or local infection;
5. Spinal cord abnormalities that require treatment;
6. Known neurological deficit (defined as motor grades < 5/5);
7. Known poor bone quality defined as T score -1.5 or less;
8. Previous spine surgery that would prevent the successful performance of the MID-C system;
9. Active systemic disease, such as AIDS, HIV, or active infection;
10. Active infection or the skin is compromised at the surgical site; and
11. Systemic disease that would affect the patient's welfare or overall outcome of the study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-20 (Estimated); Primary Completion 2028-01-20 (Estimated); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint | 5 years post MID-C system implantation
  Maintenance of major Cobb angle ≤ 30° 5 years post-surgery
Safety endpoint | 5 years post MID-C system implantation
  Serious adverse events, and device or procedure-related adverse events

IPD SHARING:
Plan to Share IPD: No